CLINICAL TRIAL: NCT00146029
Title: Companion Pharmacogenetic Study to UMCC 9900/9901
Status: Terminated | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 3-27
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Patients who participated in UMCC 9900/9901 (Phase II Studies of Tailored-Dose Docetaxel in Metastatic Breast Cancer)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose is to examine the original breast tumor material to see how much of a metabolizing enzyme (CYP3A4) is present in tumor material. The researchers want to see if this is in any way associated with how the patient responded to docetaxel. They also want to examine the genes in the tumor that are responsible for the production of CYP metabolizing enzymes, to see if they are normal or if they have polymorphisms, or change compared to 'normal' CYP metabolizing enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated on UMCC 9900/9901
* Living patients must give written informed consent

Exclusion Criteria:

* No tumor block tissue available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Anne F. Schott, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States